CLINICAL TRIAL: NCT01812538
Title: A Randomized, Single-Dose, Comparative, Positive and Placebo Controlled, Four-Way, Four Period, Cross-Over Study to Evaluate the Effect of DIC075V on QTc Intervals in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hospira, now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single
Other Study IDs: DFC-011
Record Dates: First submitted 2013-03-14; First posted 2013-03-18 (Estimated); Last update posted 2015-07-24 (Estimated); Status verified 2015-07

CONDITIONS: Ventricular Repolarization
MeSH Terms: interventions — Diclofenac

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: DIC075V
- Experimental 1 (Experimental): DIC075V 37.5 mg
  Interventions: Drug: DIC075V
- Experimental 2 (Experimental): DIC075V 75 mg
  Interventions: Drug: DIC075V
- Active control (Active Comparator): Moxifloxacin hydrochloride 400 mg
  Interventions: Drug: DIC075V

INTERVENTIONS:
Drug: DIC075V — Four single dose treatments:
  * Placebo (normal saline)
  * Moxifloxacin (positive control)
  * DIC075V 37.5 mg
  * DIC075V 75 mg
  All subjects receive each of the 4 treatments.
  Other Names: Voltaren; Voltarol; Cataflam; Zipsor

SUMMARY:
This study is conducted to evaluate the effectiveness of DIC075V on ventricular repolarization in healthy subjects compared to placebo after a single dose of DIC075V administered intravenously (IV) and to evaluate ECG assay sensitivity by evaluating the baseline-adjusted effect of a single oral (PO) moxifloxacin 400 mg dose on ventricular repolarization in healthy subjects compared to placebo. Other secondary objectives are as follows:

* To evaluate the effect of DIC075V on ventricular repolarization in healthy subjects compared to placebo at the Tmax of diclofenac and hydroxypropyl-β-cyclodextrin (HPβCD).
* To determine if there is a pharmacokinetic/pharmacodynamic (PK/PD) relationship between the duration of the QTc intervals and diclofenac and HPβCD plasma concentrations.
* Obtain additional pharmacokinetic (PK) information on diclofenac and HPβCD in healthy subjects.
* Provide additional safety information.

DETAILED DESCRIPTION:
This is a randomized, single-dose, comparative, positive and placebo controlled, 4 period, 4-way crossover study evaluating the effect of DIC075V on QTc intervals in healthy subjects. Two doses of DIC075V are tested and include moxifloxicin as a positive control and normal saline as the placebo arm. On 4 separate occasions separated by at least 72 hours, subjects are given single IV or oral (moxifloxicin) treatments. ECGs are acquired from a continuous Holter monitor and selected timepoints will be evaluated. These ECGs will be 15 seconds in duration and extracted in triplicate. Monitoring will continue for 24 hours with each treatment. The primary ECG endpoint is the baseline-adjusted QTc using the Fridericia correction (QTcF). Secondary endpoints include the baseline-adjusted QTc using the Bazett correction formula (QTcB). In addition, a population-specific regression model will be constructed with QT plotted against RR (the time elapsed between 2 consecutive R-waves). Finally, QT parameters are explored graphically in relation to PK variables Cmax, Tmax and AUC.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide signed informed consent, including Health Insurance Portability and Accountability Act (HIPAA) Authorization.
2. Healthy adult male and/or female subjects, 18-50 years of age.
3. Body mass index (BMI) between 18-30, inclusive.
4. Medically healthy with no clinically significant screening results (laboratory profiles, medical histories, ECGs, physical exam).
5. Normal blood pressure (<140 mmHg systolic and <90 mmHg diastolic).
6. Normal 12-lead ECG (QTc interval <450 millisecond (ms) for males and <470 ms for females):

   1. Consistent sinus rhythm
   2. No clinically significant conduction disorders
   3. PR interval between 120 and 230 ms
   4. HR ≤100 bpm and ≥40 bpm
   5. QRS interval ≤110 ms
   6. QT intervals that can be consistently analyzed.
7. No medical history of cardiac disease or a family history of QT prolongation.
8. No clinically significant electrolyte abnormality.
9. Subjects with a calculated creatinine clearance greater than >80 ml/min.
10. Female subjects who are of childbearing potential with a negative serum pregnancy test at Screening and at Check-in who are either sexually inactive (abstinent) for 14 days prior to Screening and throughout the study or are using two of the following acceptable birth control methods:

    * Intrauterine device (IUD) in place for at least 2 months prior to Study Day -2;
    * Barrier method (condom or diaphragm) with spermicide for at least 14 days prior to screening through study completion;
    * Hormonal contraceptive for at least 3 months prior to Study Day -2 through completion of study;
    * Surgical sterilization (vasectomy) of partner at least 6 months prior to Study Day -2.
11. Female subjects who are of non-childbearing potential with a negative serum pregnancy test at Screening and Check-in and meet at least one of the following criteria:

    * Naturally postmenopausal for a minimum of 2 consecutive years prior to Study Day -2;
    * Surgically sterile (bilateral tubal ligation with surgery at least 6 months prior to Study Day -2, hysterectomy, or bilateral oophorectomy with surgery at least 2 months prior to Study Day -2).

Exclusion Criteria:

1. History or presence of significant cardiovascular, pulmonary, hepatic, renal, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurologic, or psychiatric disease.
2. History of invasive cancer within the past 5 years (excluding non-melanoma skin cancers).
3. History of hypersensitivity or allergy to the quinolone class of antibiotics; to diclofenac or other NSAIDs; or to HPβCD or other excipients in DIC075V (monothioglycerol, sodium hydroxide, hydrochloric acid, and water for injection).
4. History or presence of alcoholism or drug abuse within the past 2 years.
5. Use of tobacco products within the previous 6 months.
6. Donation of blood within 45 days prior to Study Day -2.
7. Plasma donation within 30 days prior to Study Day -2.
8. Participation in a study of an investigational drug within 90 days prior to Study Day -2.
9. Participation in another clinical trial within 45 days prior to Study Day -2.
10. Female subjects who are pregnant or lactating.
11. Hemoglobin below the reference range for the testing laboratory.
12. Clinically significant abnormal laboratory values.
13. Abnormal ECG. The abnormality of the ECG could be a QRS duration of >110 ms, a first degree heart block defined as a PR duration >230 ms, second or third degree heart block, or a complete heart block.
14. Male subjects with a screening QTc interval ≥450 ms and female subjects with a QTc interval ≥470 ms.
15. Presence of untreated or uncontrolled blood pressure, i.e., systolic blood pressure ≥140 mmHg and/or a diastolic blood pressure ≥90 mmHg.
16. Angina, uncontrolled hypertension, clinically significant bradycardia, clinically significant cardiac arrhythmias, or any other clinically significant cardiovascular abnormality.
17. History of clinically significant syncope.
18. History of any clinically significant arrhythmias (e.g., ventricular arrhythmias, supra-ventricular arrhythmias, or atrial fibrillation).
19. History of clinically significant psychiatric illness that would prevent the subject from providing a valid Informed Consent.
20. Positive laboratory test results for hepatitis B, hepatitis C, HIV, controlled Substances, cotinine, or alcohol.
21. With the exception of hormonal contraceptives or hormone replacement therapy for females for at least 3 months piror to Study Day -2, any prescription or over-the-counter (OTC) medications, including topical medications, vitamins, herbal or dietary supplements/remedies (e.g., Saint John's Wort or Milk Thistle), within 14 days of Study Day -2.
22. With the exception of hormonal contraceptives or hormone replacement therapy for females for at least 3 months prior to Study Day -2, any planned concomitant medication for the duration of the study (except for acetaminophen up to 2 g/day).
23. History of additional risk factors for Torsade de Pointes (e.g., heart failure, hypokalemia, history of drowning survival, family history of Long QT Syndrome, family history of Short QT Syndrome, or family history of unexplainable early sudden death).
24. History of asthma attack, hives, or other allergic reactions to aspirin or other NSAID medicines.
25. History of a coronary bypass operation.
26. History of a bleeding gastric or duodenal ulcer.
27. History of skin reactions to the taking of any medications.
28. History of hepatic disorders and any symptoms associated with a hepatic disorders, e.g., nausea, tiredness, itching, flu-like symptoms, vomiting of blood, blood in the subject's bowel movements, and/or melana.
29. History of clinically significant seizures.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2009-05; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Time-matched active drug-placebo difference in baseline-adjusted QTc interval | At -1.5, -1.0, and -0.5 hours (pre-dose), and 5, 10, 15, and 30 minutes (2-min window) and 1, 2, 4, 6, 8, 12, and 23.5 hours (5-min window) on Study Days 1, 4, 7, and 10.
  The primary ECG endpoint is the time-matched active drug-placebo difference in baseline-adjusted QTc interval using the Fridericia correction formula (QTcF). The QTcF is evaluated at the time point where the maximal baseline and placebo-adjusted value is observed. These measurements are consistent with ICH E14 guidance.

SECONDARY OUTCOMES:
Time-matched active drug-placebo difference in baseline-adjusted QTc interval using the Bazett's correction formula (QTcB) evaluated at the timepoint where the maximum mean baseline- and placebo-adjusted QTcB is observed for each active treatment arm | At -1.5, -1.0, and -0.5 hours (pre-dose), and 5, 10, 15, and 30 minutes (2-min window) and 1, 2, 4, 6, 8, 12, and 23.5 hours (5-min window) on Study Days 1, 4, 7, and 10.
Time matched active drug-placebo difference in baseline adjusted QTcF at the subject-specific Tmax or the next available ECG timepoint | At -1.5, -1.0, and -0.5 hours (pre-dose), and 5, 10, 15, and 30 minutes (2-min window) and 1, 2, 4, 6, 8, 12, and 23.5 hours (5-min window) on Study Days 1, 4, 7, and 10.
Time-matched active drug-placebo difference in the maximum baseline-adjusted QTcF of each subject at each active treatment period. | At -1.5, -1.0, and -0.5 hours (pre-dose), and 5, 10, 15, and 30 minutes (2-min window) and 1, 2, 4, 6, 8, 12, and 23.5 hours (5-min window) on Study Days 1, 4, 7, and 10.

OTHER OUTCOMES:
Maximum plasma concentration (Cmax) for diclofenac and HPβCD | At Time 0 (pre-dose), and 5, 10, 15, 20, and 30 minutes and 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 18, and 23.5 hours after dosing on Study Days 1, 4, 7 and 10.
Time to Cmax (Tmax) for diclofenac and HPβCD | At Time 0 (pre-dose), and 5, 10, 15, 20, and 30 minutes and 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 18, and 23.5 hours after dosing on Study Days 1, 4, 7 and 10.
Areas under the curve to the last sample with a measurable concentration [AUC(0-t)] for diclofenac and HPβCD | At Time 0 (pre-dose), and 5, 10, 15, 20, and 30 minutes and 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 18, and 23.5 hours after dosing on Study Days 1, 4, 7 and 10.
Area under the curve from time 0 extrapolated to infinite time AUC(inf) for diclofenac and HPβCD | At Time 0 (pre-dose), and 5, 10, 15, 20, and 30 minutes and 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 18, and 23.5 hours after dosing on Study Days 1, 4, 7 and 10.
Elimination rate constant (λz) for diclofenac and HPβCD | At Time 0 (pre-dose), and 5, 10, 15, 20, and 30 minutes and 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 18, and 23.5 hours after dosing on Study Days 1, 4, 7 and 10.
Half-life (t½) for diclofenac and HPβCD | At Time 0 (pre-dose), and 5, 10, 15, 20, and 30 minutes and 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 18, and 23.5 hours after dosing on Study Days 1, 4, 7 and 10.
Total plasma clearance (CL) for diclofenac and HPβCD | At Time 0 (pre-dose), and 5, 10, 15, 20, and 30 minutes and 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 18, and 23.5 hours after dosing on Study Days 1, 4, 7 and 10.
Volume of distribution (Vz) for diclofenac and HPβCD | At Time 0 (pre-dose), and 5, 10, 15, 20, and 30 minutes and 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 18, and 23.5 hours after dosing on Study Days 1, 4, 7 and 10.

CONTACTS AND LOCATIONS:
Locations (1):
- Cetero Research, Fargo, North Dakota, United States

REFERENCES:
- [Derived] Carr DB, McDonnell Moorehead T, Bouchard A, Sprenger CR, Hamilton DA, Lang E, Madden D, Lacouture PG, Wright C 4th. Effects of injectable HPbetaCD-diclofenac on the human delayed rectifier potassium channel current in vitro and on proarrhythmic QTc in vivo. Clin Ther. 2013 May;35(5):646-58. doi: 10.1016/j.clinthera.2013.03.014. Epub 2013 Apr 8. PMID 23578606